CLINICAL TRIAL: NCT00106210
Title: Early Detection, Intervention, and Neurobiology in Autism: Early Intervention Portion
Brief Title: School- and Home-Based Early Intervention for Toddlers With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Rebecca Landa, Director of the Center for Autism and Related Disorders (CARD) and Professor, Johns Hopkins University School of Medicine, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U54MH066417 (NIH); U54MH066417 (NIH); DDTR BD-DD
Record Dates: First submitted 2005-03-21; First posted 2005-03-22 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-07

CONDITIONS: Autistic Disorder; Autism
Keywords: Child
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Behavioral Intervention (experimental)
  Interventions: Behavioral: Early intervention blending several tx approaches, w/ focus
- 2 (Active Comparator): Behavioral Intervention 2
  Interventions: Behavioral: Early intervention blending several treatment approaches

INTERVENTIONS:
Behavioral: Early intervention blending several tx approaches, w/ focus — Early intervention blending several different treatment approaches, with a focus on certain skills
  Arms: 1
Behavioral: Early intervention blending several treatment approaches — Early intervention blending several different treatment approaches
  Arms: 2

SUMMARY:
This study will determine the impact of early intervention on the communication and social development of toddlers with autism.

DETAILED DESCRIPTION:
Autism is a condition that affects brain development, often leading to difficulties in social, emotional, and educational functioning. This study will determine whether early intervention can improve such functioning in toddlers with autism.

Each treatment session will last 6 months. Children with an autism spectrum disorder will be enrolled in one of two parallel classes and will receive one of two treatments 4 days a week for the duration of the session. Children in each class will receive the same amount and level of intervention, but with a different goal focus. Treatments will be school- and home-based; parents will receive instruction on administering the at-home part of the treatment. The intervention will include environmental engineering, developmental approaches, adaptations of traditional behavioral approaches, and contemporary behavioral approaches that apply principles of applied behavior analysis in more naturalistic teaching frameworks. A series of measures including scales, interviews, and observations will be used to assess the children at baseline, study completion, and 6 months after study completion. The children will be videotaped during the school-based intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autism spectrum disorder
* Parent or guardian willing to give informed consent for child's participation
* Developmental level above 9 months on the Visual Reception Scale of the Mullen Scales of Early Learning and on the Adaptive Behavior Composite of the Vineland Adaptive Behavior Scales
* English is primary language for child and family

Exclusion Criteria:

* Evidence of vision or hearing impairment
* Diagnosis of fragile X syndrome, Rett syndrome, tuberous sclerosis, neurofibromatosis, phenylketonuria, or congenital rubella
* History of severe birth trauma or traumatic brain injury
* Siblings with autism spectrum disorder

Ages: 18 Months to 33 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2003-05; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Receptive language skills | Pre-tx, Post-tx, and 6 month follow up
Expressive language skills | Pre-tx, Post-tx, and 6 month follow up

SECONDARY OUTCOMES:
Social cognitive skills | Pre-tx, Post-tx, and 6 month follow up
Social emotional functioning | Pre-tx, Post-tx, and 6 month follow up
Play skills | Pre-tx, Post-tx, and 6 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Landa, PhD, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Landa RJ, Holman KC, O'Neill AH, Stuart EA. Intervention targeting development of socially synchronous engagement in toddlers with autism spectrum disorder: a randomized controlled trial. J Child Psychol Psychiatry. 2011 Jan;52(1):13-21. doi: 10.1111/j.1469-7610.2010.02288.x. Epub 2010 Dec 3. PMID 21126245
- See also: Click here for the Center for Autism and Related Disorders (CARD) at the Kennedy Krieger Institute Web site — http://www.kennedykrieger.org/kki_cp.jsp?pid=1394
- See also: Click here for the Autism and Neuro-Psychiatric Disorders Research at the Kennedy Krieger Institute Web site — http://www.kennedykrieger.org/kki_research.jsp?pid=1800